CLINICAL TRIAL: NCT01698268
Title: The Efficacy of Transverse Abdominis Plane (TAP) Block in Children Undergoing Hydrocelectomy and/or Hernia Repair
Brief Title: Study of Transverse Abdominis Plane (TAP) Block in Children Undergoing Hydrocelectomy and/or Hernia Repair Surgery
Acronym: TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaveh Aslani, MD (Other)
Responsible Party: Sponsor-Investigator, Kaveh Aslani, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-213
Record Dates: First submitted 2012-08-14; First posted 2012-10-02 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Hydrocele; Inguinal Hernia
MeSH Terms: conditions — Testicular Hydrocele; Hernia, Inguinal | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP Group (Experimental): Enrolled subjects will receive a TAP block with 0.5cc/kg of 0.25% ropivacaine.
  Interventions: Procedure: TAP block
- Local Infiltration Group (Active Comparator): Enrolled subjects will receive will receive local infiltration of 0.5 cc/kg of 0.25% ropivacaine.
  Interventions: Procedure: Local Infiltration

INTERVENTIONS:
Procedure: TAP block — TAP Block will be performed under ultrasound guidance via Sonosite device with an in-plane technique by the anesthesiologist.
  Arms: TAP Group
Procedure: Local Infiltration — Local infiltration of 0.5 cc/kg of 0.25% ropivacaine will be administered by the surgeon.
  Arms: Local Infiltration Group

SUMMARY:
Study measures the difference in pain after hernia &/or hydrocele repair based on site of local anesthesia injection.

DETAILED DESCRIPTION:
This single-center, prospective, single blind, randomized study will enroll up to 50 subjects who are scheduled for elective hydrocelectomy and/or hernia repair. At Beaumont Health System, post-operative pain management in children is managed either via oral/parenteral opiates and opiate adjuncts, surgeon-administered field blocks (instillation of local anesthetics in the general area of incision), or via regional techniques (spinal, epidural, or peripheral nerve blocks). We have designed this study to determine if there is improved qualitative and quantitative post-operative pain control in patients receiving TAP block versus intraoperative peri-incisional, surgeon administered field block. Once informed consent has been given, each patient will be randomized (like flip of the coin) to either Transverse Abdominis Plane Block (TAP Block)or surgeon administered anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Children 2-8 years of age
* Elective inguinal hernia repair, inguinal hernia repair with peritoneoscopy and/or hydrocelectomy to be performed in the Center for Children's Surgery, Beaumont Hospital, Royal Oak
* American Society of Anesthesiologists physical status classification 1 and 2 (patients that have either no systemic illness, or mild systemic disease that is well controlled, eg. mild asthma)

Exclusion Criteria:

* History of allergy to study medications
* Enrollment in concurrent research study
* Pregnant patients*
* Students/trainees/staff*
* Mentally disabled/cognitively impaired*

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaveh Aslani, MD, Principal Investigator — Beaumont Health
Locations (1):
- Beaumont Health System, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-center, prospective, single blind, randomized study enrolled subjects who were scheduled for elective hydrocelectomy and/or hernia repair at Beaumont Hospital-Royal Oak. The first procedure was on 3/16/2012 and the last one was on 11/12/2014.
Period: Overall Study
Arm/Group | TAP Group | Local Infiltration Group
Started | 25 | 25
Completed | 23 | 24
Not Completed | 2 | 1
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: Data not included for patients removed from study by physician
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP Group | Local Infiltration Group | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 24 | 47
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 20 | 21 | 41
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: FLACC: Face, Legs, Activity, Cry, and Consolability Pain Assessment Scale (FLACC)
Description: FLACC: Face, Legs, Activity, Cry, and Consolability Pain Assessment Scale (FLACC), a five-item, three point scale that measures pain behavior on a scale of 0 - 2 which are summed to result in a total score of 0 - 10. Clinical judgment is used to interpret pain. The higher the score on the FLACC correlates with a higher pain score (0= no behaviors indicative of pain and 10= five behaviors indicative of significant pain). This scale was evaluated by blinded post-operative anesthesia care unit (PACU) Registered Nurses (RNs) at admission to PACU.
Time Frame: Admission into PACU
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | TAP Group | Local Infiltration Group
Number analyzed (Participants) | 23 | 24
units on a scale | 0 [0 to 0] | 0 [0 to 3.5]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of consent through the time of a followup phone call 24 hours post discharge from the hospital.
Arm/Group | TAP Group | Local Infiltration Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 9/23 | 7/24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAP Group (N=23) | Local Infiltration Group (N=24)
Agitation (General disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Restlessness (General disorders) | 0 (0) | 1 (1)
Incisional pain (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
skin inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Of the 47 treated patients, the local infiltration was administered by 8 different surgeons while the TAP block was administered by 2 different anesthesiologists.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No